CLINICAL TRIAL: NCT02957487
Title: Maxillary 3-implant Removable Prostheses Without Palatal Coverage on Locator Abutments - a Prospective Cohort Study
Brief Title: Maxillary 3-implant Removable Prostheses Without Palatal Coverage on Locator Abutments
Status: Completed | Type: Observational
Sponsor: University of Tromso (Other)
Responsible Party: Sponsor
Other Study IDs: REK 2013/1446
Record Dates: First submitted 2016-10-21; First posted 2016-11-07 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-04

CONDITIONS: Edentulous Maxilla

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Denture supported by 3 dental implants — Metal-reinforced denture without palatal coverage incorporating nylon rings retained by friction to Locator abutments fitted on top of dental implants

SUMMARY:
The aims of this clinical study conducted at a dental specialty clinic in Drammen, Norway are to assess the clinical outcomes of patients with an edentate upper jaw having been treated with a removable full prosthesis supported by 3 implants to restore function and aesthetics. Clinical variables beyond implant dimensions and intraoral location, such as recall routines, maintenance needs, patient satisfaction and quality of life, will also be appraised and contrasted with an aim to elucidate their association with clinical outcomes. Specific evaluation will be done with regard to the following outcome criteria:

* crestal bone levels and periodontal conditions around implants
* incidence rates of biological, technical, traumatic failures / complications related to implants
* incidence rates of biological, technical, mechanical, esthetic failures/complications with prosthesis and prosthetic components A secondary objective is to identify the different risk factors for biological failures / complications, including the influence of medical conditions and tobacco use.

DETAILED DESCRIPTION:
Materials and Methods The protocol is submitted to the Research Ethics Board of the Northern Norway in order to obtain ethics approval prior to commencing the study. All patients will obtain an invitation letter detailing the objectives of the study and requested to sign a consent letter prior to clinical examinations according to principles for good research practice. All patients will be offered a free implant hygiene session and prosthesis cleaning.

Study population All patients treated in a private dental clinic in Drammen, Norway having received a maxillary removable full prosthesis supported on 3 dental implants will be invited to attend evaluations of their intra-oral status annually after implant installation and solicited about treatment satisfaction and daily oral functions. These patients were initially not offered maintenance care at the completion of their treatment.

The implants that have been used are made from titanium with a microrough surface (Astra Tech Implant System, Dentsply Implants, Mølndal, Sweden). All implants have been placed according to the manufacturer's instructions (http://www.dentsplyimplants.no/nb-NO/Implantatsystem/Prosedyrer/Treatment-planning) and fitted with precision attachments (Locator, ZEST Anchors, Escondido, CA, USA. The removable prostheses were made from heat cured poly-methyl-metacrylate (PMMA) incorporating three active matrices).

Recall Procedure Each patient will be invited by letter followed up by a phone call to attend an examination visit. The patients will complete a questionnaire related to changes in general health aspects, their experiences and satisfaction with the reconstructions and eventual need for repair sessions during the last year. Specifically, the medical history and the smoking history (e.g. pack/years) will be assessed. Recordings will be made of general and local factors which may affect the prognosis of the implants and prosthesis. This includes the occurrence of systemic disease since implant placement, regular medication used by patients, smoking status, dental treatment received since implant placement, recall frequency at the dental hygienist and the last dental examination appointment.

Collection of Data from Patients' Charts

General information will be gathered from the patients' charts. Patients' age, self-reported smoking habits and the number of cigarettes per day, medical history, medication intake, reason for tooth loss and the date of prosthesis insertion will be recorded in "patient's summary forms". Type and distribution of implants will be retrieved from patients' charts. Cases with a chart documentation of an incidence of biological or mechanical complications during the follow-up period will be closely reviewed and recorded as following:

1. History of implant loss (Biological complication):

   Period of service before failure is traced in months for each lost implant. Lost implants will be categorized in three groups: 1) "Early Failure" which refers to implants lost before the insertion of the definite prosthesis. 2) "One-year Failure" addressing implants failed within the first year of loading. 3) "Late Failure" including implants lost more than one year following the insertion of the final prosthesis (Roos-Jansåker et al 2006).
2. History of peri-implant mucositis or peri-implantitis (biological complication):

   Any recorded incidence of inflammation and suppuration related to the gingival tissue surrounding implants in patients' charts will be gathered and transferred to "patients' summary forms".
3. History of various technical problems encountered following the insertion of the removable prosthesis (mechanical complications):

Any history of mechanical complications such as attachment loosening/fracture and incidences of cracks, chippings and fractures in resin teeth, acrylic body and prosthesis will be recorded in "patients' summary forms".

Post-operation peri-apical radiographs, taken at the day of "stage-one" surgery, will be retrieved from patient's charts and used as the reference point of supporting bone level for each implant. Reference bone levels on mesial and distal sides are determined by measuring the distance between implant platform and the most apical point of the alveolar crestal bone surrounding implant. A mean value between the mesial and distal sides is used for each implant as the reference marginal bone level.

ELIGIBILITY:
Inclusion Criteria:

Edentulous maxilla Competence to sign the informed consent form describing the study

Exclusion Criteria:

Lack of jaw bone for the placement of dental implants without the need for bone regeneration.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated in a private dental clinic in Drammen, Norway
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Intra-oral status | 3 years
  The radiographic examination will comprise periapical radiographs or an orthopantomogram. The clinical examination include a basic periodontal examination with the use of an UNC-15 (University of North Carolina) manual periodontal probe. Outcomes measured will be presence or absence of peri-implant suppuration or fistula, the modified plaque and sulcus bleeding indices) and the probing depths.
Condition of prosthesis and implants | 3 years
  The removable prosthesis will be examined for any technical flaws. Adverse technical events include loss of retention, or fracture and/or chipping of the removable prosthesis. Adverse mechanical events include loosening of the male attachment or fracture of an implant. The stability of all implants will be assessed, and any sign of mobility along with pain and discomfort will be interpreted as a definitive sign of implant failure.

SECONDARY OUTCOMES:
Implant bone level changes | 3 years
  Reference bone levels on the mesial and distal sides will be measured relative to baseline measurements made at the time of delivery of denture
Patient-reported satisfaction outcome | 5 years
  A self-reported Denture Satisfaction Scale questionnaire (Allen et al. 2001).
Patient-reported quality of life outcome | 5 years
  The short form version of the Oral Health Impact Profile questionnaire (OHIP-20) (Allen & Locker 2002).

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn Jokstad, DDS, PhD, Principal Investigator — UiT The Arctic University of Norway
Locations (1):
- Tannlege Arild Mo, Drammen, Norway

REFERENCES:
- [Background] Mo A, Hjortsjo C, Olsen-Bergem H, Jokstad A. Maxillary 3-implant removable prostheses without palatal coverage on Locator abutments - a case series. Clin Oral Implants Res. 2016 Oct;27(10):1193-1199. doi: 10.1111/clr.12724. Epub 2015 Nov 14. PMID 26566604